CLINICAL TRIAL: NCT05268848
Title: Foot Thermography With the Use of Different Plantar Orthosis Lining Materials
Brief Title: Thermography of the Foot With Plantar Orthosis Liners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Elena Escamilla Martinez, Assistant proffesor. Nursing Department., Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Termografiaforros2022
Record Dates: First submitted 2021-12-22; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Foot Orthosis; Temperature
Keywords: infrared thermography; orthopodia; thermometry

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Termography PRE (Experimental): Foot thermography before lining test
  Interventions: Other: Thermographic photo
- Termography POST (Experimental): Foot thermography after wearing 2 types of liner for three hours (one on each foot)
  Interventions: Other: Thermographic photo
- Thermographic comparations (Active Comparator): Thermographic comparations between PRE and POST measurements
  Interventions: Other: Thermographic photo

INTERVENTIONS:
Other: Thermographic photo — Barefoot patient, thermographic photo of the sole of the feet is taken

SUMMARY:
Objetive: To analyze the thermal effects of the types of liners used in the manufacture of the foot orthoses, as well as to establish the thermal differences among them.

Design: Quantitative, experimental, longitudinal and prospective study. Subjects: 47 individuals selected randomly, over 20 years of age Methods: 4 types of liner were studied: natural skin, synthetic leather, perforated E.V.A and E.V.A. without perforation.

ELIGIBILITY:
Inclusion Criteria:

People wearing sanitary footwear. 20-35 years Not having smoked or taken alcohol or exciting drinks before evaluation Without cream on the sking and not being exposed to UV rays.

Exclusion Criteria:

young or old people with respect to the age of study smokers or drinkers

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Foot temperature measurement PRE | for a month
  The camera Flir E60BX was used, placed on a tripod one meter away from the feet. A photo of the sole of the foot was taken.

SECONDARY OUTCOMES:
Foot temperature measurement POST | for a month
  Photo after the use of linings inside the shoe

OTHER OUTCOMES:
Foot temperature measurment by area | for 3 months
  Using the Flir Tools software, 3 areas were selected on each foot, calculating the average temperature in each area: metatarsal heads, lateral region and heel center.

CONTACTS AND LOCATIONS:
Overall Officials: ELENA ESCAMILLA MARTÍNEZ, Principal Investigator — University of Extremadura
Locations (1):
- Elena Escamilla Martínez, Plasencia, Cáceres, Spain